CLINICAL TRIAL: NCT01550445
Title: Prospective Controlled Protocol for 3 Months Steroid Withdrawal With Tacrolimus, Basiliximab, and Mycophenolate Mofetil in Renal Transplant Recipients
Brief Title: Steroid Withdrawal Immunosuppression After Renal Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Chang kwon oh, Professor, Department of Surgery, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-CRO-08-067
Record Dates: First submitted 2012-02-15; First posted 2012-03-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Steroid withdrawal, Kidney transplantation
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- steroid withdrawal (No Intervention): The clinical outcome after kidney transplantation, under the immunosuppression of steroid withdrawal starting at 3 months post-transplantation using tacrolimus, mycophenolate mofetil, and basilixumab should be analyzed.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Those patients who fulfill the entry criteria enter in this prospective controlled trial of steroid withdrawal starting at three months after transplantation

SUMMARY:
The investigators analyze the clinical outcome of steroid withdrawal protocol starting at 3 months after kidney transplantation using tacrolimus, Mycophenolate Mofetil (MMF), and basiliximab. This study is an open-label, prospective, controlled clinical trial in a single center. Those patients who fulfill the entry criteria could enter in this prospective controlled trial of steroid withdrawal three months after transplantation.

DETAILED DESCRIPTION:
Those patients who fulfill the entry criteria enter in this prospective controlled trial of steroid withdrawal starting at three months after transplantation. The entry criteria include 1) no episode of clinically treated nor biopsy confirmed acute rejection up to entry; 2) serum creatinine level equal to or less than 2 mg/mL on three separate measurements; 3) no proteinuria (urine protein less than 1000 mg/24 hours; 4) tacrolimus trough level > 5 ng/ml without signs of nephrotoxicity; 5) agreement to follow the study protocol.

For the patients who enter into the protocol, prednisolone would be slowly withdrawn by 2.5 mg in every two weeks until 8 weeks after entering the protocol (5 months post-transplantation). The patients visit every week, and they are closely monitored with symptoms and signs, blood cell count, chemistry, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 13 years who received a primary kidney transplant
* Subject who is using CNI ± purine synthesis inhibitor + steroid without change within the past 3 months (except the dosage)
* serum creatinine < 2 mg/dL and the variation of serum creatinine < 30% during the past 3 months
* Proteinuria ≤ 1g quantified by 24 hour urine or spot urine protein/creatinine ratio < 1.0
* Subjects who agree with written informed consent

Exclusion Criteria:

* Subjects who received combined non-renal transplantation.
* Subject who received re-transplantation
* Deceased donor without a heartbeat
* Patients with hypersensitivity to Mycophenolate sodium, Mycophenolate acid or Mycophenolate Mofetil or to any of the excipients.
* Patient with HGPRT(Hypoxanthin e-guanine phosphoribosyl-transferase) such as Lesch-Nyhan syndrome and kelley-Seegmiller syndrome.
* HLA-identical living related donor
* ABO blood group incompatible
* HIV, HBsAg, or HCV Ab tests (+)
* Abnormal liver function test (AST or ALT or total bilirubin> upper normal limit x3) ANC < 1,500/μL or WBC < 2,500/μL or platelet < 750,000/μL
* Women who are either pregnant, lactating, planning to become pregnant in the next 12 months.
* Subjects with history of cancer, except successfully treated, localized nonmelanocytic skin cancer Subjects with clinically significant infections within the past 3 months.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
the incidence of biopsy-confirmed acute rejection. | 12 months
  The primary efficacy variable was the incidence of biopsy-confirmed acute rejection.

SECONDARY OUTCOMES:
death, graft loss | 12 months
  The secondary efficacy variables included the cumulative incidence of a composite endpoint of death, and graft loss;
adverse events and serious adverse events | 6 months , 12 months
  The proportion of successfully steroid-withdrawn and steroid-free population at 6 months and at 12 months post-transplantation as well as the safety variables including the incidence of adverse events and serious adverse events, [blood pressure, lipid levels (total cholesterol), BUN (blood urea nitrogen) and blood glucose levels]

CONTACTS AND LOCATIONS:
Overall Officials: Chang kwon oh, M.D.,Ph. D., Principal Investigator — Department of surgery, Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea

REFERENCES:
- [Derived] Oh CK, Kim SJ, Kim JH, Lee JH. Prospective controlled protocol for three months steroid withdrawal with tacrolimus, basiliximab, and mycophenolate mofetil in renal transplant recipients. J Korean Med Sci. 2012 Apr;27(4):337-42. doi: 10.3346/jkms.2012.27.4.337. Epub 2012 Mar 21. PMID 22468094